CLINICAL TRIAL: NCT05298826
Title: Recombinant Factor VII for the Conservative Management Trials of Intractable Postpartum Haemorrhage: is it a Drug Effect , Operator Experience or Inherent Result of the Aetiology.
Brief Title: Recombinant Factor VII for Intractable Postpartum Haemorrhage
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Recombinant factor VII
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior staff has started the management and called for the senior staff.
  Interventions: Drug: recombinant factor VIIa
- senior staff. managed the case from the start
  Interventions: Drug: recombinant factor VIIa

INTERVENTIONS:
Drug: recombinant factor VIIa — using recombinant factor VIIa

SUMMARY:
Postpartum haemorrhage remains at the top of the causes of maternal deaths in both developed and developing countries .

DETAILED DESCRIPTION:
Major postpartum haemorrhage is a dangerous complication that accounts for the highest maternal morbidity rate

ELIGIBILITY:
Inclusion Criteria:

* Women with severe resistant postpartum hemorage

Exclusion Criteria:

* women without postpartum hemorage

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with resistant postpartum hemorage
Study Population: women who has resistant postpartum hemorage
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
The number of women who had hysterectomy | 24 hours
  number of women resistant to the treatment and needed hysterectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Doaaa Alaa, Cairo, Egypt